CLINICAL TRIAL: NCT05758220
Title: Magnetic Resonance Imaging of the Brain in Children With Autism Spectrum Disorder (ASD)
Brief Title: MRI Brain (Volumetry, fMRI & MRS) in Autism
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed AbuDeif Sayed, Radio-Diagnosis & Interventional Radiology Specialist, Assiut University
Other Study IDs: MRI Brain in Autism
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder
Keywords: MRI brain in ASD
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — Structural MRI volumetry, resting functional MRI & MR spectroscopy

SUMMARY:
To reach a feasible method for diagnosing Autism Spectrum Disorder (ASD) outcome measures:

1. Primary (main):

   Measurement of various brain structures, including the total brain volume, the volumes of specific brain regions (such as the amygdala, hippocampus, and cerebellum), and the thickness of the cortex.

   Detection of other concurrent lesions, e.g. tuberous sclerosis
2. Secondary (subsidiary):

levels of various neurotransmitters, such as glutamate and GABA, and other metabolites, such as N-acetyl aspartate (NAA), in specific regions of the brain Assessing neural activity and connectivity in the brain in the resting state

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a heterogeneous disorder (or collection of related disorders) of multifactorial etiology, and with a great range in severity of symptoms. ASD affects approximately 1 in 166 children and is four times more prevalent in boys than in girls. Core features of individuals with autism include 1) impairment in reciprocal social interactions; 2) verbal and nonverbal communication deficits; 3) repetitive and ritualized behaviors; and 4) a narrow range of interests. Approximately 30% of individuals with ASD manifest some degree of mental retardation.

Magnetic-resonance (MR) examination allows researchers and clinicians to noninvasively examine brain anatomy in vivo. Structural MR examination is widely used to investigate brain morphology because of its high contrast sensitivity and spatial resolution, and because it entails no radiation exposure; the last feature is particularly important for children and adolescents.

Functional magnetic resonance imaging (fMRI) has proven to be a useful tool to investigate aberrant neurobiological function in ASDs because of its excellent contrast properties, spatial resolution, and temporal resolution. fMRI uses specialized pulse sequences to localize metabolic correlates of neural activity linked to relevant neurocognitive processes

Investigating brain network activity during the resting state has emerged as a new method that eliminates the caveats of task-based fMRI studies

The fMRI signal is measured during the resting state and the data is analyzed based on a connectivity approach between subdivisions. To date, brain network activity during the resting state has been investigated in subjects with ASD and typical development in numerous studies. Overall, intrinsic connectivity between subdivisions of the brain is altered in patients with ASD compared to controls.

MRS's finding is that gamma oscillations are reduced in ASD patients. Gamma oscillations are generated by GABAergic neurons and are involved in sensory binding and higher cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Children clinically diagnosed with Autism Spectrum Disorder.
* Males and Females.
* Children with an IQ of more than 70%

Exclusion Criteria:

* Severe forms of ASD.
* Children with IQ less than 70%.
* Children with claustrophobia.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with Autism Spectrum Disorder
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Structural MRI brain volumetry | Baseline
  Measurement of various brain structures, including the total brain volume, the volumes of specific brain regions (such as the amygdala, hippocampus, and the cerebellum), and the thickness of the cortex.

SECONDARY OUTCOMES:
resting functional MRI & MR spectroscopy | Baseline
  levels of various neurotransmitters, such as glutamate and GABA, and other metabolites, such as N-acetyl aspartate (NAA), in specific regions of the brain Assessing neural activity and connectivity in the brain in the resting state

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed ab AbdelTawab, MD, Study Chair — Assiut University

REFERENCES:
- [Result] Chakrabarti S, Fombonne E. Pervasive developmental disorders in preschool children. JAMA. 2001 Jun 27;285(24):3093-9. doi: 10.1001/jama.285.24.3093. PMID 11427137
- [Result] Eliez S, Reiss AL. MRI neuroimaging of childhood psychiatric disorders: a selective review. J Child Psychol Psychiatry. 2000 Sep;41(6):679-94. PMID 11039681
- [Result] Chao HT, Chen H, Samaco RC, Xue M, Chahrour M, Yoo J, Neul JL, Gong S, Lu HC, Heintz N, Ekker M, Rubenstein JL, Noebels JL, Rosenmund C, Zoghbi HY. Dysfunction in GABA signalling mediates autism-like stereotypies and Rett syndrome phenotypes. Nature. 2010 Nov 11;468(7321):263-9. doi: 10.1038/nature09582. PMID 21068835